CLINICAL TRIAL: NCT04577001
Title: Letrozole in Patients With Hepatopulmonary Syndrome: A Double-Blind Randomized Clinical Trial
Brief Title: Letrozole in Patients With Hepatopulmonary Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Recruitment Numbers
Sponsor: Mayo Clinic (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Hilary M. DuBrock, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-005779
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Hepatopulmonary Syndrome
MeSH Terms: conditions — Hepatopulmonary Syndrome | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letrozole Group (Experimental): Subjects with hepatopulmonary syndrome will get the study drug letrozole
  Interventions: Drug: Letrozole
- Placebo Group (Placebo Comparator): Subjects with hepatopulmonary syndrome will get the study placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Letrozole — 2.5 mg orally daily for 6 months
  Arms: Letrozole Group
Drug: Placebo — No active ingredient taken orally daily for 6 months
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to assess the safety, tolerability and possible benefit of letrozole compared to placebo in patients with Hepatopulmonary Syndrome.

DETAILED DESCRIPTION:
This study is a phase II randomized, double-blind, placebo-controlled parallel trial of 20 subjects with hepatopulmonary syndrome designed to assess the effect of letrozole 2.5 mg orally daily or placebo for 6 months on the alveolar-arterial oxygen gradient (AaPO2).

Subjects at each site will be screened at outpatient clinic visit appointments and interested qualified subjects will be consented and offered participation in this trial. Once consent has been obtained baseline values will be established and subjects will begin letrozole with follow-up clinic visits and testing at 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of moderate to very severe hepatopulmonary syndrome which consists of having all 3 of the following conditions:

  * Presence of liver disease or portal hypertension
  * Intrapulmonary shunting on contrast-enhanced echocardiogram
  * Hypoxemia [A-a gradient ≥15mmHg (or ≥20mmHg if age >64) and PaO2<80mmHg on arterial blood gas testing]
* Child-Pugh class A or B liver disease
* MELD score < 20
* ≥ 18 years old
* Female subjects must be post-menopausal (defined as 12 months of spontaneous amenorrhea or 6 weeks postsurgical bilateral oophorectomy without or without hysterectomy)
* Ability to provide informed consent

Exclusion Criteria

* Enrollment in a clinical trial or concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 28 days of baseline
* Current hepatic encephalopathy
* Expectation of liver transplant within six months of randomization
* Concomitant lung disease defined as restriction (TLC < 70%) or obstruction (FEV1 < 80% & FEV1/FVC < 70%)
* Inability to comply with the study protocol
* Osteoporosis
* Premenopausal women (those who have not reached 1 year absence of menarche)
* Vulnerable study population, including imprisoned individuals, or those who cannot consent on their own.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary M DuBrock, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Letrozole Group | Placebo Group
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Subject became ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study terminated due to low recruitment numbers. No subjects were enrolled in the Letrozole group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole Group | Placebo Group | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Alveolar-Arterial Oxygen
Description: To determine whether letrozole affects alveolar-arterial oxygen gradient (AaPO2) at 6 months in patients with HPS.
Time Frame: 6 months
Population: Study terminated due to low recruitment numbers. Data was not collected on the one enrolled participant for this outcome measure due to withdrawal after becoming ineligible prior to outcome measure timeframe completion.
Arm/Group | Letrozole Group | Placebo Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Hormone Levels
Description: To determine whether letrozole affects estradiol, progesterone, testosterone levels at 6 months
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Letrozole Group | Placebo Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Oxygen Saturation
Description: To determine whether letrozole affects oxygen saturation from pulse oximetry at 3 months 6 months and distance walked in 6 minutes in patients with HPS
Time Frame: 3 and 6 months
Population: as for outcome 1
Arm/Group | Letrozole Group | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Side Effects
Description: To determine the safety and adverse effects associated with letrozole administration in patients with HPS
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Letrozole Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of 37 days.
Description: Study terminated due to low recruitment numbers. No subjects were enrolled in the Letrozole group.
Arm/Group | Letrozole Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Terminated study due to low recruitment numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT04577001/Prot_SAP_000.pdf